CLINICAL TRIAL: NCT03145818
Title: Evaluation of Veteran Directed Home and Community Based Services
Brief Title: Evaluation of Veteran-Directed Home and Community Based Services
Acronym: VD-HCBS Eval
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SDR 16-194; NCT04795791 (obsolete NCT alias)
Record Dates: First submitted 2017-05-01; First posted 2017-05-09 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Functional Impairment; Caregiving
Keywords: dissemination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Veterans: Veterans will be the primary group for whom the VD-HCBS Program is implemented. Veterans enrolled in VD-HCBS will be functionally impaired
  Interventions: Other: VD-HCBS
- Caregivers: Caregivers support Veterans independence in their home and community
  Interventions: Other: VD-HCBS
- VHA Coordinators: VHA VD-HCBS Coordinators allow the program to operate within the VA
  Interventions: Other: VD-HCBS
- ADNA Coordinators: ADNA Coordinators engage with the Veteran, Caregivers, and VA Coordinators to ensure the Veteran is able to maintain independence
  Interventions: Other: VD-HCBS

INTERVENTIONS:
Other: VD-HCBS — Like the participant-directed programs developed for Medicaid programs,VD-HCBS maximizes Veteran-centered care and independence. VD-HCBS provides Veterans with a monthly financial allotment based on an assessment of the extent of their need for assistance with personal care due to injury or the impact of disease

SUMMARY:
Veteran-Directed Home and Community Based Services (VD-HCBS) is focused on preserving Veteran's independence and the VA Office of Geriatrics and Extended Care is planning an expansion of VD-HCBS to 90 additional VA Medical Centers over the next 3 years. This proposal seeks to evaluate the VD-HCBS expansion to capture comprehensive information on the impact of VD-HCBS on Veterans' and Caregivers' outcomes, as well as, to identify how the program was implemented.

DETAILED DESCRIPTION:
In the next decade, there will be a doubling of older Veterans for whom the VA has a requirement to provide long-term care. At a cost of $110,000 per year for long-term care, Geriatrics and Extended Care (GEC) is seeking to preserve Veteran independence in the community. VD-HCBS is a person-centered consumer-directed program that provides Veterans the opportunity to self-direct their long-term services and supports (LTSS) and continue to live independently at home. GEC is planning to expand VD-HCBS to an additional 90 VAMCs over the next 3 years. This proposal will provide important outcomes and context to the VD-HCBS expansion. The specific aims of this proposal are: Aim 1: To describe the impact of VD-HCBS on Veterans' satisfaction, unmet need for services, quality of life and independence using mixed methods. Aim 1 will utilize operations data to describe the change in Veteran-reported satisfaction, unmet needs, and independence from enrollment in VD-HCBS to 3 and 12 months. Additionally, the investigators will conduct interviews with Veterans to capture their experiences with the program. Aim 2: To understand the effect of VD-HCBS on Caregivers' well-being. Aim 2 will compare Caregivers' financial strain, depressive symptoms, caregiving stress, and health status and positive caregiver experiences to a propensity matched population from existing VA data to determine the impact of the VD-HCBS program on Caregivers. Aim 3: To examine the implementation of the VD-HCBS program expansion. Aim 3 will utilize the Consolidated Framework for Implementation Research and Expert Recommendations for Implementing Change to interview coordinators, and other key informants, from VA and ADNA VD-HCBS pairs. The analysis will shed light on how contextual factors and implementation strategies relate to implementation and Veteran outcomes. VD-HCBS has tremendous opportunity to improve the fiscal outlook of GEC's LTSS while delivering the highest level of Veteran-centered care. In concert with the outcomes of VD-HCBS, this implementation evaluation will be critical to determining how the VA system, in partnership with community-based organizations, implements programs and illuminating important leverage points to facilitate implementation effectiveness. With the diverse team assembled and the comprehensive evaluation proposed, the investigators will produce evidence to inform VA program implementation and dissemination, a critical component of the VA's priorities to develop high-performing, highly-reliable, and consistent networks.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who are eligible and enrolled in VD-HCBS at the expansion VAMCs

Exclusion Criteria:

* Non-Veterans
* Those not eligible or enrolled in VD-HCBS
* Enrolled in VD-HCBS at a non-expansion VAMC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans enrolled in VD-HCBS tend to be older with functional impairments which could precipitate facility based care placement
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L. Rudolph, MD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (2):
- United States (2):
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garrido MM, Allman RM, Pizer SD, Rudolph JL, Thomas KS, Sperber NR, Van Houtven CH, Frakt AB. Innovation in a Learning Health Care System: Veteran-Directed Home- and Community-Based Services. J Am Geriatr Soc. 2017 Nov;65(11):2446-2451. doi: 10.1111/jgs.15053. Epub 2017 Aug 21. PMID 28832927
- See also: VA VD-HCBS — https://www.va.gov/GERIATRICS/Guide/LongTermCare/Veteran-Directed_Care.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment letters to Veterans, Caregivers and Coordinators were sent inviting them to participate in qualitative interviews.
Groups:
- Veterans: Veterans will be the primary group for whom the VD-HCBS Program is implemented. Veterans enrolled in VD-HCBS will be functionally impaired. The surveys are given at the onset of the program and quarterly and yearly thereafter.
  VD-HCBS: Like the participant-directed programs developed for Medicaid programs,VD-HCBS maximizes Veteran-centered care and independence. VD-HCBS provides Veterans with a monthly financial allotment based on an assessment of the extent of their need for assistance with personal care due to injury or the impact of disease
Period: Overall Study
Arm/Group | Veterans | Caregivers | VHA Coordinators | ADNA Coordinators
Started | 99 | 8 | 10 | 9
Completed | 8 | 0 | 10 | 9
Not Completed | 91 | 8 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Veterans enrolled in the VD-HCBS program completed a life satisfaction survey on unmet needs, satisfaction and quality of life. Caregivers completed a well-being survey focusing on financial strain, depressive symptoms, caregiving stress, health status and positive caregiver experiences.
Groups:
- Total: Total of all reporting groups
Arm/Group | Veterans | Caregivers | VHA Coordinators | ADNA Coordinators | Total
Number analyzed (Participants) | 99 | 8 | 10 | 9 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age information was not collected from coordinators.
  years
    number analyzed (Participants) | 99 | 8 | 0 | 0 | 107
    (all) | 75.4 (13.6) | 63 (12.0) |  |  | 74.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender information was not collected for coordinators.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity information was not collected for coordinators.
  Participants
    number analyzed (Participants) | 99 | 8 | 0 | 0 | 107
    Hispanic or Latino | 0 | 0 |  |  | 0
    Not Hispanic or Latino | 99 | 8 |  |  | 107
    Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race information was not collected for coordinators.
  Participants
    number analyzed (Participants) | 99 | 8 | 0 | 0 | 107
    American Indian or Alaska Native | 3 | 0 |  |  | 3
    Asian | 0 | 0 |  |  | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Black or African American | 37 | 1 |  |  | 38
    White | 52 | 6 |  |  | 58
    More than one race | 1 | 0 |  |  | 1
    Unknown or Not Reported | 6 | 1 |  |  | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 99 | 8 | 10 | 9 | 126

OUTCOME MEASURES:

1. Primary Outcome: Veteran's Unmet Need for Services, Satisfaction, Unmet Needs, and Quality of Life.
Description: Satisfaction Survey Number of Veterans responding to VA-specific program survey questions on Veteran satisfaction, unmet needs, and quality of life. Veterans were asked to respond to a 6 question survey by choosing a number from a scale (either from 1-10 or 1-5; low numbers typically indicating satisfaction; higher numbers indicating dissatisfaction) to indicate their level of overall satisfaction with their current health needs and ability to participate in daily activities.
Time Frame: 12 months
Population: Veterans enrolled in the Veteran Directed Home and Community Based Services program.
  Six Veterans did not participate in the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Veterans
Number analyzed (Participants) | 93
Participants
  1. Satisfaction of VA home services | 71
  2. Need additional help with everyday activities | 63
  3. Able to attend recreational/social activities | 35
  4. Worry about being able to remain in home | 39
  5. Enough choice for services and products | 66
  6. General life satisfaction | 60

2. Primary Outcome: Caregiver Well-being Survey
Description: Number of caregivers who responded to a VA specific Caregiver survey on financial strain, depressive symptoms, caregiving stress, and health status and positive caregiver experiences. Caregivers were asked to choose the best answer from a scale that reflected the level of intensity (low numbers typically indicating less intensity than the higher numbers) of common caregiving stressors.
Time Frame: 9 months
Population: Caregivers who participated in a caregiver well-being survey.
Measure: Count of Participants; unit: Participants
Groups:
- Caregivers: Caregivers supporting Veterans independence in their home and community
  VD-HCBS: Like the participant-directed programs developed for Medicaid programs,VD-HCBS maximizes Veteran-centered care and independence. VD-HCBS provides Veterans with a monthly financial allotment based on an assessment of the extent of their need for assistance with personal care due to injury or the impact of disease
Arm/Group | Caregivers
Number analyzed (Participants) | 8
Participants
  Serious Economic Situation | 4
  Stressed between caregiving and other responsibili | 3
  Reported Poor Health | 0
  Felt lonely or isolated | 5

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Veterans: Veterans enrolled in VD-HCBS have needs for services, the primary outcome are the needs which are not currently met
- Caregivers: Caregiving wellbeing will be measured with a composite of financial strain, depressive symptoms, caregiving stress, and health status and positive caregiver experiences.
- VA Coordinators; VHA Coordinators: This semi-structured interview will identify constructs from the Consolidated Framework for Implementation Research and the Expert Recommendations for Implementing Change (ERIC).
Arm/Group | Veterans | Caregivers | VA Coordinators | VHA Coordinators
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/8 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/8 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/99 | 0/8 | 0/10 | 0/9

LIMITATIONS AND CAVEATS:
Unexpected events slowed expansion of VD-HCBS

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT03145818/Prot_SAP_000.pdf